CLINICAL TRIAL: NCT01449981
Title: Development and Testing of Adolescent Twelve-Step Facilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John F. Kelly, Associate Director MGH Center for Addiction Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA R01AA019664
Record Dates: First submitted 2011-10-04; First posted 2011-10-10 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Alcohol Abuse; Alcohol Dependence; Drug Abuse; Drug Dependence
Keywords: Adolescents; Alcohol Abuse; Alcohol Dependence; Drug Abuse; Drug Dependence; Substance Use Disorder; Alcoholics Anonymous; Motivational Enhancement Therapy; Cognitive Behavioral Therapy
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated Twelve-Step Facilitation (Experimental)
  Interventions: Behavioral: Integrated Twelve-Step Facilitation
- Cognitive Behavioral Therapy (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Integrated Twelve-Step Facilitation — The iTSF condition will include review of treatment goals and overall review of progress, coping skills, real life practices, emotions/mood management, how to make changes in one's social network and discussions about how 12-step meetings can be helpful in one's recovery efforts. In addition, speakers from 12-step fellowships such as Alcoholics Anonymous (AA) and Narcotics Anonymous (NA) will be invited to share their experiences and discuss myths and facts related to attendance at 12-step meetings as well as answer any questions participants have about these fellowships.
  Other Names: iTSF
  Arms: Integrated Twelve-Step Facilitation
Behavioral: Cognitive Behavioral Therapy — The CBT condition will include review of progress, coping skills, group exercises, real life practice, and emotions/mood management.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy

SUMMARY:
This study is the first to develop and test in a randomized experimental design the efficacy of an integrated 12-step facilitation intervention tailored for young people. In the first phase of the study, the investigators are developing and revising a preliminary manual for the two sessions individually-delivered Motivational Enhancement Therapy (MET) component and subsequent 8 session group-delivered Cognitive-Behavioral Therapy (CBT) component which will integrate Twelve-step Facilitation (TSF). Forty adolescents each will complete the preliminary integrated TSF protocol. In the second phase of the study, the investigators will compare integrated TSF (iTSF) to standard treatment (MET/CBT) in a randomized experimental design for adolescent substance use disorder with 60 adolescents. As a result, the investigators will examine potential mechanisms that may underlie the efficacy of iTSF in improving alcohol and other drug use outcomes. The investigators will test group differences on potential mechanisms of change (e.g., Alcoholics Anonymous/Narcotics Anonymous attendance and involvement) and whether these variables are associated with substance use outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Young people between the ages of 14 and 21 that meet criteria for alcohol or other drug abuse or dependence.

Exclusion Criteria: Youth

* with an active psychotic disorders
* who are in another substance use disorder (SUD) treatment program or receiving SUD related psychotherapy that could conflict with our treatment
* with a history of severe or complicated withdrawal (e.g., alcohol seizure history)
* who may be using alcohol/drugs prior to study entry at levels likely to result in severe withdrawal complications, in the absence of any history
* taking addiction treatment medications (e.g., Buprenorphine)
* who cannot speak English because the treatment and assessment instruments will be conducted in English

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Percent Days Abstinent (PDA) | Up to 9 months
  Given the goals of both treatments will be abstinence, the main outcome analyses and effect size estimates will be based upon biochemically verified 90 day point-prevalence of PDA. These will be captured using Form-90 (Miller & Del Boca, 1994) which will be used to examine substance use (including number of days used and first and last dates of use within the time period), as well as other treatment experiences in the past 90 days.

SECONDARY OUTCOMES:
Treatment Acceptability | Up to 3 months
  Participants will also complete weekly treatment feedback measures to inform the treatment manual.

CONTACTS AND LOCATIONS:
Overall Officials: John F. Kelly, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Center for Addiction Medicine 60 Staniford Street, Boston, Massachusetts, United States